CLINICAL TRIAL: NCT06450392
Title: The Effect of Local and Systemic Tranexamic Acid on Edema and Ecchymosis in Orbital Surgery - a Prospective, Multicenter, Randomized, Double-blinded, Control Trial
Brief Title: The Effect of Local and Systemic Tranexamic Acid on Edema and Ecchymosis in Orbital Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-15945
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Orbital Edema; Orbital Ecchymosis
Keywords: Orbital Surgery
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, double-blinded, controlled trial. On the day of surgery in the preoperative suite, study participants will be randomly allocated to one of three groups via computer-generated random numbers as described in the Arms and Interventions section.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: IV TXA (Experimental): 1g intravenous tranexamic acid (Pfizer, New York, NY) 20 minutes prior to surgery
  Interventions: Drug: Tranexamic Acid in NaCl,Iso-Os 1,000 Mg/100 mL (10 Mg/mL) INTRAVEN INTRAVENOUS SOLUTION, PIGGYBACK (ML); Drug: normal saline - injection
- Group 2: Local TXA (Experimental): 1-2mL of subcutaneous tranexamic acid 100 mg/mL (manufactured concentration, Pfizer, New York, NY) mixed with local anesthetic to the orbit two minutes prior to incision
  Interventions: Drug: Tranexamic acid injection; Drug: normal saline - intravenous
- Group 3: Control (Placebo Comparator): Normal saline and subcutaneous local anesthetic to both eyelids (i.e. standard procedure) as control group
  Interventions: Drug: normal saline - injection; Drug: normal saline - intravenous

INTERVENTIONS:
Drug: Tranexamic acid injection — 100 mg/mL (manufactured concentration) local TXA injection in the orbit
  Arms: Group 2: Local TXA
Drug: Tranexamic Acid in NaCl,Iso-Os 1,000 Mg/100 mL (10 Mg/mL) INTRAVEN INTRAVENOUS SOLUTION, PIGGYBACK (ML) — 1g IV TXA
  Arms: Group 1: IV TXA
Drug: normal saline - injection — 0.9% Normal Saline injection in the orbit
  Arms: Group 1: IV TXA; Group 3: Control
Drug: normal saline - intravenous — 0.9% IV Normal Saline
  Arms: Group 2: Local TXA; Group 3: Control

SUMMARY:
Tranexamic acid (TXA) is a synthetic reversible competitive inhibitor to plasminogen lysine receptor, which prevents plasmin formation and stabilizes the fibrin matrix, thus reducing bleeding. While recent studies have demonstrated the antifibrinolytic benefits of TXA in obstetric and gynecologic conditions, traumatic hemorrhage, cardiac surgery, total knee arthroplasty, and more, there is a paucity of clinical data on TXA use in plastic surgery. The aim of this study is to evaluate the effect of local and systemic TXA on postoperative periocular ecchymosis/edema in orbital surgery.

DETAILED DESCRIPTION:
Patients, who will be undergoing orbital surgery anyways, will be given the option to participate in the study. Informed consent will be obtained in clinic during the preoperative consultation. On the day of surgery in the preoperative suite, study participants will be randomly allocated to one of three groups via computer-generated random numbers:

Group 1: will receive 1g intravenous tranexamic acid (Pfizer, New York, NY) 20 minutes prior to surgery. Group 2: will receive 1.7 mL of subcutaneous tranexamic acid 100 mg/mL (Pfizer, New York, NY) with local anesthetic to the orbit two minutes prior to incision. Group 3: will receive intravenous normal saline and subcutaneous local anesthetic (i.e. standard procedure) as control group.

Twenty minutes before incision time, all patients will receive an intravenous solution. This will be either saline (placebo, participants in group 2 and 3) or 1g of tranexamic acid (participants in group 1). All operations will be performed using the standard of care technique and surgical instruments. All surgery will be performed under intravenous sedation with local anesthesia. Standard skin marking will be drawn, then the surgeon will inject each patient subcutaneously with either (1) a 5 cc mixture of TXA (100 mg/mL) mixed with 2% lidocaine with epinephrine and 0.5% marcaine with epinephrine in a 1:1:1 ratio (local TXA, Group 2) or (2) normal saline 0.9% sodium chloride mixed with 2% lidocaine with epinephrine and 0.5% marcaine with epinephrine in a 1:1:1 ratio (Group 1, Group 3). Degree of ecchymosis and edema in the postoperative photographs will be assessed separately by two graders. Graders will be blinded to treatment groups, and the photos will be completely deidentified.

Immediately following the procedure, the surgeon will take standardized photographs. The surgeon will also take standardized photographs at the regular 7-day postoperative visit. These photos will be deidentified and analyzed for degree of ecchymosis and edema by two blinded graders who will rate the photos using a standard five point grading scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = profound) as described in the respective outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orbital surgery (decompressions, fracture repairs, enucleations, eviscerations, etc.)
* Patients who are at least 18 years of age
* Patients that have the capacity to consent

Exclusion Criteria:

* Any history of previous orbital surgery
* Any patient undergoing multiple simultaneous periocular surgical procedures
* Any patient with active infection
* History of stroke or seizure
* History of bleeding/clotting disorder
* Patients who do not comply with the required postoperative follow-up schedule
* Patients who are allergic to tranexamic acid
* Patients who have taken anticoagulant/antiplatelet agents (including aspirin) within 7 days prior to surgery
* Patients who have periocular ecchymosis or edema prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Degree of Ecchymosis | 0 days and 7 days postoperatively
  Degree of ecchymosis on postoperative day zero (POD0) and postoperative day 7 (POD7) as graded on a 5 point Likert scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = profound) by two independent graders. The two scores will be averaged for inclusion in analysis. Scores will be aggregated to calculate means and standard deviations (SDs) for each group. Higher scores are associated with increased severity of ecchymosis.
Degree of Edema | 0 days and 7 days postoperatively
  Degree of edema on postoperative day zero (POD0) and postoperative day 7 (POD7) as graded on a 5 point Likert scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = profound) by two independent graders. The two scores will be averaged for inclusion in analysis. Scores will be aggregated to calculate means and standard deviations (SDs) for each group. Higher scores are associated with increased severity of edema.

SECONDARY OUTCOMES:
Patient Satisfaction with edema | 7 days postoperatively
  Patients asked how satisfied they are with their edema postoperatively. Responses will be scored as 0 (not satisfied at all), 1 (somewhat unsatisfied), 2 (neutral), 3 (somewhat satisfied), or 4 (completely satisfied). Responses will be summed and mean scores and standard deviations (SDs) will be reported for each group. Higher scores correlate with increased degree of satisfaction.
Patient Satisfaction with ecchymosis | 7 days postoperatively
  Patients asked how satisfied they are with their ecchymosis postoperatively. Responses will be scored as 0 (not satisfied at all), 1 (somewhat unsatisfied), 2 (neutral), 3 (somewhat satisfied), or 4 (completely satisfied). Responses will be summed and mean scores and standard deviations (SDs) will be reported for each group. Higher scores correlate with increased degree of satisfaction.
Other side effects | 7 days postoperatively
  Patients will be asked if they had any seizure, focal weakness, lower extremity pain, difficulty breathing, chest pain, or any emergency room visit (to assess for adverse effects including thromboembolic event or seizure). Responses will be recorded as either "Thromboembolic event occurred" or "Thromboembolic event did not occur." Seizure events will be recorded in the same way. The number of patients with thromboembolic events and/or seizures will be summarized by the study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Barmettler, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kono S, Lee PAL, Kakizaki H, Takahashi Y. Orbital haematoma after orbital fracture repair using silicone, polytetrafluorethylene, and poly-L-lactic acid/hydroxyapatite implants. Br J Oral Maxillofac Surg. 2021 Nov;59(9):1036-1039. doi: 10.1016/j.bjoms.2021.01.002. Epub 2021 Jan 15. PMID 34531075
- [Background] Colomina MJ, Contreras L, Guilabert P, Koo M, M Ndez E, Sabate A. Clinical use of tranexamic acid: evidences and controversies. Braz J Anesthesiol. 2022 Nov-Dec;72(6):795-812. doi: 10.1016/j.bjane.2021.08.022. Epub 2021 Oct 7. PMID 34626756
- [Background] Paramo R, Cheng T, Malik A, Fan J, Barmettler A. Effect of Tranexamic Acid on Intra- and Postoperative Bleeding in Eyelid Surgery: A Prospective, Randomized, Multicenter, Double-Masked, Control Trial. Ophthalmic Plast Reconstr Surg. 2024 May-Jun 01;40(3):331-335. doi: 10.1097/IOP.0000000000002583. Epub 2024 Apr 12. PMID 38624153
- [Background] Marous CL, Farhat OJ, Cefalu M, Rothschild MI, Alapati S, Wladis EJ. Effects of Preoperative Intravenous Versus Subcutaneous Tranexamic Acid on Postoperative Periorbital Ecchymosis and Edema Following Upper Eyelid Blepharoplasty: A Prospective, Randomized, Double-Blinded, Placebo-Controlled, Comparative Study. Ophthalmic Plast Reconstr Surg. 2024 Sep-Oct 01;40(5):523-532. doi: 10.1097/IOP.0000000000002633. Epub 2024 Apr 29. PMID 38687303
- [Background] Artymowicz, A., & Shinder, R. (2022). Effect of subcutaneous tranexamic acid on hemostasis and ecchymosis in dacryocystorhinostomy: A double-blind, placebo-controlled, randomized clinical trial. Poster session presented at the ASOPRS 2022 Conference, Chicago, IL, United States.
- [Background] Zilinsky I, Barazani TB, Shenkman B, Weisman O, Farber N, Martinowitz U. Topical Hemostatic-Anesthetic Solution to Reduce Bleeding During Mohs Micrographic Surgery: A Case Control Study. J Drugs Dermatol. 2016 Jul 1;15(7):851-5. PMID 27391635
- [Background] Horrow JC, Van Riper DF, Strong MD, Grunewald KE, Parmet JL. The dose-response relationship of tranexamic acid. Anesthesiology. 1995 Feb;82(2):383-92. doi: 10.1097/00000542-199502000-00009. PMID 7856897
- [Background] Schroeder RJ 2nd, Langsdon PR. Effect of Local Tranexamic Acid on Hemostasis in Rhytidectomy. Facial Plast Surg Aesthet Med. 2020 May/Jun;22(3):195-199. doi: 10.1089/fpsam.2020.0061. Epub 2020 Mar 31. PMID 32228311